CLINICAL TRIAL: NCT02053415
Title: Study of the Effect of Krill Oil Supplement on Omega-3 Fatty Acid Index and Tolerance
Brief Title: Krill Oil as Supplementation to Healthy Young Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Olympic Seafood AS (Industry)
Responsible Party: Principal Investigator, Bodil Bjørndal, Researcher, University of Bergen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Krill oil pilot-2014
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: krill oil; omega-3 index; plasma lipid profile; tolerance; young adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Krill oil low dose (Experimental): 3 capsules krill oil per day, for 28 days
  Interventions: Dietary Supplement: Krill oil low dose
- Krill oil high dose (Experimental): 9 capsules krill oil per day, for 28 days
  Interventions: Dietary Supplement: Krill oil high dose

INTERVENTIONS:
Dietary Supplement: Krill oil low dose — 3 capsules krill oil per day
  Other Names: Rimfrost Sublime krill oil
  Arms: Krill oil low dose
Dietary Supplement: Krill oil high dose — 9 capsules krill oil per day
  Other Names: Rimfrost Sublime krill oil
  Arms: Krill oil high dose

SUMMARY:
The purpose of this study is to examine whether 4 weeks daily intake of krill oil can change the omega-3 index (content of the long chained fatty acids EPA and DHA in relation to the total fatty acids) in the membrane in red blood cells. We investigate this at two different doses. Furthermore, the purpose of the study is also to examine the effect of the krill oil intake on plasma lipids (triacylglycerol, phospholipids and cholesterol), plasma fatty acid composition, as well as product tolerance in healthy, young individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults

Exclusion Criteria:

* Disease/illness
* Not able to swallow supplements in capsule form
* Not willing to take blood samples

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Fatty acid composition in red blood cells (the membrane) | Day 0 (baseline), and day 28 (end)
  Change in fatty acid composition and omega-3 index (sum of % EPA and DHA)

SECONDARY OUTCOMES:
Fasting plasma lipid status | Day o (baseline), and day 28 (end)
  * Change in triacylglycerol levels.
  * Change in phospholipid levels.
  * Change in cholesterol levels (total, ester, free, HDL, LDL).
Fatty acid composition in plasma. | Day 0 (baseline), and day 28 (end)
  Change in fatty acid composition and omega-3 index (sum of % EPA and DHA).
Fasting glucose and glucose tolerance. | Day 0 (baseline), and day 28 (end)
  Change in fasting glucose and glucose tolerance.
Tolerance of and compliance with intervention | Day 28 (end)
  Questionnaire-based

CONTACTS AND LOCATIONS:
Overall Officials: Per Bakke, Professor, Principal Investigator — University of Bergen
Locations (1):
- Department of Clinical Science, University of Bergen, Bergen, Bergen, Norway